CLINICAL TRIAL: NCT03874741
Title: A Phase II Study of Evaluating Recombinant Human Anti-EGFR Monoclonal Antibody (SCT200) and Standard Chemotherapy for Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: SCT200 Plus Platinum-based Chemotherapy in Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT200-B202
Record Dates: First submitted 2019-03-08; First posted 2019-03-14 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck Cancer; Epidermal growth factor receptor; SCT200
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm - Experimental (Experimental): Anti-EGFR monoclonal antibody DDP(75mg/m2),d1; 5-FU(750mg/m2),d1-5, every 21d; PF chemothrapy up to 6 cycles. 6.0mg/kg of SCT200 will be administered once a week for a maximum of 6 cycles. After 6 cycles, 8.0mg/kg of SCT200 will be administered every two weeks until disease progression.
  Interventions: Drug: SCT200

INTERVENTIONS:
Drug: SCT200 — Anti-EGFR monoclonal antibody DDP(75mg/m2),d1; 5-FU(750mg/m2),d1-5, every 21d; PF chemothrapy up to 6 cycles. 6.0mg/kg of SCT200 will be administered once a week for a maximum of 6 cycles. After 6 cycles, 8.0mg/kg of SCT200 will be administered every two weeks until disease progression
  Other Names:
  • SCT200
  Other Names: Anti-EGFR monoclonal antibody

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of first-line with recombinant anti-EGFR monoclonal antibody#SCT200#and standard chemotherapy in patients with Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma.

DETAILED DESCRIPTION:
This open label, single-arm and multicenter phase II study is designed to evaluate Objective Response Rate (ORR) of first-line with anti-EGFR monoclonal antibody#SCT200#and standard chemotherapy in Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this clinical trial and sign an informed consent form;
* Male or female, age ≥ 18 and ≤ 75 years old;
* ECOG fitness status score 0 to 1;
* Recurrent and/or metastatic HNSCC (except nasopharyngeal carcinoma) diagnosed by pathology #
* Not suitable for topical treatment. Patients with only recurrent disease (no metastasis) must have received radiotherapy (as post-operative adjuvant therapy or as a treatment for locally advanced HNSCC) as a "localized area treatment" and radiotherapy must be completed at least 6 months prior to screening imaging#
* Laboratory inspection:
* Blood routine: neutrophils ≥1.5×l09/L, platelets≥75×109/L, hemoglobin≥80g/L;
* Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST), ALT and AST ≤ upper limit of normal value × 3 for liver metastasis, ALT and AST ≤ upper limit of normal value for liver metastases × 5; total bilirubin ( TBIL) ≤ upper limit of normal value × 2.0;
* Renal function: creatinine (Cr) ≤ normal upper limit × 1.5;
* Electrolyte: Magnesium ≥ normal lower limit;
* According to the RECIST standard version 1.1, there is at least one measurable tumor lesion.

Exclusion Criteria:

* Patients with a history of central nervous system metastasis or a history of central nervous system metastasis before screening. For patients with clinically suspected central nervous system metastasis, imaging confirmation must be performed within 28 days prior to enrollment to exclude central nervous system metastasis;
* Received systemic chemotherapy for advanced or metastatic HNSCC, but do not include induction chemotherapy, concurrent chemoradiotherapy or adjuvant chemotherapy (the end of this treatment must be more than 6 months from the first trial);
* There are other medical history of malignant tumors, except that the malignant lesions have been treated with therapeutic measures 5 years or more before enrollment and there are no known active lesions. The investigator judges that the risk of recurrence is low; Non-melanoma skin cancer, and no evidence of worsening disease; adequately treated cervical cancer in situ, and no evidence of worsening disease; prostatic intraepithelial neoplasia, no evidence of prostate cancer recurrence;
* known to be allergic to antibodies or other components contained in the test drug;
* have received EGFR antibodies (such as panitumumab, cetuximab or its analogs), or small molecule EGFR inhibitors (such as gefitinib, erlotinib, lapatinib, etc.);
* In the 4 weeks or 4 weeks before enrollment, they received anti-tumor drugs (such as chemotherapy, hormone therapy, immunotherapy, antibody therapy, radiotherapy, etc.) or received research drug treatment and could not be included in the evaluation by the investigator. Pain-free palliative radiotherapy for bones;
* At the time of enrollment, patients still had ≥2 peripheral neuropathy or hearing loss;
* Patients have been enrolled in other study devices or study drug studies at screening time, or have been deactivated for less than or equal to 4 weeks from other study drugs or study devices;
* Conduct or plan major surgery within 4 weeks prior to enrollment;
* Received transfusion, erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GMCSF) within 2 weeks prior to enrollment;
* Clinically significant cardiovascular disease (defined as: unstable angina, symptomatic congestive heart failure (New York Heart Association [NYHA]

  ≥ II), uncontrollable severe arrhythmia);
* Myocardial infarction occurred within 6 months prior to enrollment;
* History of interstitial lung disease (ILD), such as interstitial pneumonia, pulmonary fibrosis, or evidence of ILD on baseline chest CT or MRI;
* have clinical symptoms, require clinical intervention or serous effusion (such as pleural effusion and ascites) with a stabilization time of less than 4 weeks;
* medical or psychiatric history or laboratory abnormal medical history that may interfere with the interpretation of the results;
* Patients who are pregnant or breast-feeding, or who plan to be pregnant during the treatment period and within 6 months after the end of treatment;
* Patients (including male or female patients) who are unwilling to receive effective contraception during the treatment period and within 6 months after the end of treatment;
* HCV antibody positive; or HIV positive; or HBV test results: HBsAg positive and / or HBcAb positive and HBV DNA ≥ 104 copy number or ≥ 2000 IU / ml;
* Patients have active or uncontrollable infections (except for simple urinary tract infections or upper respiratory tract infections) requiring systemic treatment within 2 weeks or 2 weeks prior to enrollment;
* known patients have alcohol or drug addiction;
* The investigator believes that patients have other conditions that may affect their adherence to protocol adherence and study indicators, and are not suitable for patients participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 year
  ORR is defined as proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 during trial treatment.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 1 year
  The achievement of any stable disease#SD#, partial response (PR) or complete response (CR), according to RECIST v1.1 criteria.
Progresssion free survival(PFS) | 1 year
  PFS is defined as the time from first dose of SCT200 until the date of first documentation of progression or date of death, whichever occurs first,according to RECIST v1.1 criteria.
Overall survival(OS) | 1 year
  OS is defined as time from first dose of SCT200 until the date of death from any cause
Immunogenicity | 1 year
  Serum anti-SCT200 antibody levels before and after administration
EORTC QLQ-C30 | 1 year
  Median scores for each item and domain will be reported at each time point. 30 items questionnaire with answers ranging from 1=not at all to 4=very much includes five functional scales (physical, role, emotional, cognitive and social), three symptom scales (fatigue, nausea & vomiting and pain) and a global health status/QOL scale.
  Furthermore, it contains six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties)
EORTC QLQ-H&N35 | 1 year
  European organization for research and treatment of cancer quality of life questionnaire head and neck 35(EORTC QLQ-H & N 35) is a specific questionnaire developed by the European Organisation for Research and Treatment of Cancer for head and neck cancer. The module includes 35 questions Assessing symptoms and side effects of treatment, social function and body image/sexuality .This scale includes seven symptoms subscales that measure pain, swallowing, senses problems, speech problems, trouble with social eating, trouble with social Contact, and less sexuality, and also has 11 subscales related with teeth, opening mouth, dry mouth, sticky saliva, coughing, ill feeling, weight loss, weight gain, use of painkillers, nutritional supplements, and feeding tubes. Standardize the original scores, with scores ranging from 0 to 100, with higher scores representing more serious problems.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital Chinese academy of medical sciences, Beijing, Beijing Municipality, China